CLINICAL TRIAL: NCT02386345
Title: EU Focal Impulse and Rotor Modulation Registry -Topera E-FIRM Registry-
Brief Title: Topera E-FIRM Registry
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Collaborators: I-Med-Pro GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: E-FIRM 02
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Atrial Fibrillation
Keywords: FIRM procedure
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a registry to assess the safety and effectiveness of FIRM guided procedures for the treatment of symptomatic any type of atrial fibrillation.

FIRM (Focal Impulse and Rotor Modulation) guided ablation is defined as ablating rotors identified by the FIRMap® basket catheter for visualising of rotors with the RhythmView® mapping system. In addition to the FIRM guided ablation any other ablation method could be applied.The acute success of FIRM ablations is defined as elimination of rotors defined by absence of rotors.

Data items will be collected, if available, consistent and applicable with routine and standard clinical care at each participating site.

DETAILED DESCRIPTION:
Prospective and retrospective enrollment is possible.

ELIGIBILITY:
Inclusion Criteria:

reported incidence of at least 2 documented episodes of symptomatic AF (paroxysmal, persistent or long standing persistent) during the 3 months preceding the initial AF ablation attempt of at least one Class I or III anti-arrhythmia drug with failure defined as recurrence of symptomatic AF or adverse drug effect resulting in stopping medication

Exclusion Criteria:

women who are pregnant

As this is a registry only data of patients will be included who have been treated according to the current AF guidelines.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who are receiving a FIRM guided AF ablation and are selected in accordance with the current AF guidelines are eligible for the participation in the registry
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2015-03; Primary Completion 2017-05-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, Prof. Dr., Principal Investigator — Herzzentrum Leipzig - Universitätsklinik; Kristin Ruffner, PhD, Study Director — Abbott
Locations (9):
- Germany (8):
  - Städtisches Klinikum Karlsruhe GmbH, Karlsruhe, Baden-Würtemberg
  - Herz- und Gefäßklinik, Bad Neustadt an der Saale, Bavaria
  - Klinikum Coburg GmbH, Coburg, Bavaria
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci, Potsdam, Brandenburg
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia
  - Zentrum für klinische Prüfungen in der Facharztzentrum Dresden-Neustadt GbR, Dresden, Saxony
  - Herzzentrum Leipzig, Leipzig, Saxony
  - Unfallkrankenhaus Berlin, Berlin
- Erasmus Medical Center, Rotterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Registry Population: All patients enrolled in the registry
Period: Overall Study
Arm/Group | Registry Population
Started | 299
Completed | 197
Not Completed | 102
Not completed — Not treated | 14
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 5
Not completed — Repeat Procedure | 10
Not completed — Did not complete 12-month follow-up | 72

BASELINE CHARACTERISTICS:
Arm/Group | Registry Population
Number analyzed (Participants) | 299
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 204
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (4.9)
New York Heart Association Class [Count of Participants; unit: Participants] — The New York Heart Association Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity; the limitations/symptoms are in regard to normal breathing and varying degrees in shortness of breath and/or angina.
  Class I = no limitation of physical activity. Class II = slight limitation Class III = marked limitation Class IV = unable to carry on any physical activity without discomfort
  Participants
    Class I | 94
    Class II | 79
    Class III | 37
    Not reported | 89
Type of Atrial Fibrillation [Count of Participants; unit: Participants]
  Paroxysmal | 38
  Persistent | 248
  Long lasting | 11
  Not reported | 2
Left Ventricle Ejection Fraction [Mean (Standard Deviation); unit: percent] | 55.8 (8.5)
Left Atrium Diamter [Mean (Standard Deviation); unit: millimeter] | 47.2 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Success
Description: Acute Success was defined as the elimination (by ablation) of all identified rotors
Time Frame: day of procedure
Measure: Count of Participants; unit: Participants
Groups:
- Analysis Population: All treated patients
Arm/Group | Analysis Population
Number analyzed (Participants) | 285
Participants | 165

2. Primary Outcome: Number of Participants With 12-Month Success
Description: Single procedure freedom from atrial fibrillation recurrence
Time Frame: 12-months after index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Population
Number analyzed (Participants) | 242
Participants | 101

3. Primary Outcome: Number of Participants With Acute Safety Success
Description: Acute safety success was defined as freedom from Serious Adverse Events at 7 days after index procedure
Time Frame: 7 days after index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Population
Number analyzed (Participants) | 271
Participants | 257

4. Primary Outcome: Number of Participants With 12-Month Safety Success
Description: Success was defined as freedom from Serious Adverse Events at 12-months after index procedure
Time Frame: 12-months after index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Population
Number analyzed (Participants) | 218
Participants | 184

5. Other Pre Specified Outcome: Number of Participants With 6-Month Safety Success
Description: Success was defined as freedom from Serious Adverse Events at 6-months after index procedure
Time Frame: 6-months after index procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Analysis Population
Number analyzed (Participants) | 256
Participants | 232

ADVERSE EVENTS:
Time Frame: 12-months
Arm/Group | Registry Population
All-Cause Mortality (participants affected / at risk) | 0/299
Serious Adverse Events (participants affected / at risk) | 34/299
Other Adverse Events (participants affected / at risk) | 0/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Registry Population (N=299)
Recurrent Atrial Fibrillation (Cardiac disorders) | 9 (13)
Bleeding with medical intervention (Vascular disorders) | 7 (8)
Pericardial effusion (Vascular disorders) | 2 (2)
Atrioesophageal fistula (Cardiac disorders) | 1 (1)
Transient ischemic attack (Cardiac disorders) | 3 (3)
Stroke (Vascular disorders) | 1 (1)
Cardiac Resynchronization Therapy Pacemaker implantation (Surgical and medical procedures) | 2 (2)
Cavotricuspid isthmus ablation (Surgical and medical procedures) | 2 (2)
Dyspnea (Vascular disorders) | 1 (1)
Heart rhythm disorder (Cardiac disorders) | 1 (2)
High position right hemotoma (Vascular disorders) | 1 (1)
Intramuscular hemorrhage (Vascular disorders) | 1 (1)
Lip laceration (Surgical and medical procedures) | 1 (1)
Non-sustained ventricular tachycardia (Cardiac disorders) | 1 (1)
Pacemaker implantation (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All manuscripts should be submitted to the sponsor for review and comment prior to submission to the publisher.

DOCUMENTS (1):
  • Study Protocol (2014-07-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT02386345/Prot_000.pdf